CLINICAL TRIAL: NCT03197454
Title: Brain Enhancement Training Towards Elders Resilience to Aging (BETTER Aging)
Brief Title: Brain Enhancement Training Towards Elders Resilience to Aging
Acronym: BETTER Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Posit Science Corporation (Industry)
Collaborators: University of Iowa (Other); The University of Texas at Dallas (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSC-0605-17
Record Dates: First submitted 2017-06-21; First posted 2017-06-23 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Age-related Cognitive Decline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Treatment (Experimental): Computerized plasticity-based adaptive cognitive training requiring a total maximum of 50 treatment sessions, up to 5 sessions per week, 42 minutes per session.
  Interventions: Other: Computerized Plasticity-Based Adaptive Cognitive Training
- Active Comparator (Active Comparator): Commercially available computerized training requiring a total maximum of 50 treatment sessions, up to 5 sessions per week, 42 minutes per session.
  Interventions: Other: Commercially available computerized training

INTERVENTIONS:
Other: Computerized Plasticity-Based Adaptive Cognitive Training — Forty-two minutes of training on computerized exercises that targets processing speed, memory and attention.
  Arms: Experimental Treatment
Other: Commercially available computerized training — Forty-two minutes of training on computerized, casual video games.
  Arms: Active Comparator

SUMMARY:
This study is a parallel arm, double-blind, randomized, controlled clinical trial to assess the efficacy of an experimental software program designed to improve cognitive functions versus a computer-based software control. Both the study and the software being investigated meet the criteria of Non-Significant Risk.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the effects of the experimental treatment (cognitive training) further outlined in this protocol on the cognitive abilities (e.g., processing speed, attention, working memory, and executive function), brain functionality, functional status and quality of life of individuals with age-related cognitive decline as compared to a computer-based active control.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 65 years of age or older
* Participant must be a fluent English speaker
* Participant must have adequate sensorimotor capacity to perform the program, including visual capacity adequate to read from a computer screen at a normal viewing distance, auditory capacity adequate to understand normal speech, and motor capacity adequate to control a computer mouse
* Participant must not have evidence of dementia as indicated by the Montreal Cognitive Assessment (MoCA)

Exclusion Criteria:

* Participant with any medical illnesses, injuries or conditions predisposing to imminent functional and/or cognitive decline
* Participant requiring caregiver assistance in dressing/personal hygiene
* Participant with severe visual deficits (including visual neglect, partial field cuts, anopias) and/or severe hearing deficit that would prevent use of the computerized treatment program
* Participant with recent participation of computer-delivered cognitive training within 2 years of consent
* Participant with claustrophobia or any other contraindication to MRI scanning
* Participant with inability to complete a 1-hour MRI
* Pregnant women
* Participant with any implanted devices above the waist (e.g., cardiac pacemaker or auto-defibrillators, neural pacemaker, aneurysm clips, cochlear implant, metallic bodies in the eye or central nervous system, any form of wires or metal devices that may concentrate radio frequency fields)
* Participants with active suicidal ideation with specific plan and intent or suicide-related behaviors within 2 months of consent as measured by the Columbia-Suicide Severity Rating Scale (C-SSRS)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 147 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2021-07-16 (Actual)

PRIMARY OUTCOMES:
Change in performance on global cognitive composite score | At 3 months and at 9 months
  Change in performance on global cognitive composite score based on the average of all normalized assessment measures.

SECONDARY OUTCOMES:
Change in performance on processing speed composite score | At 3 months and at 9 months
  Change in performance on processing speed will be measured using the composite score created by averaging the z-scores of Pattern Comparison, Letter Comparison, and Digit Symbol Coding tasks.
Change in performance on memory | At 3 months and at 9 months
  Change in performance on memory will be measured using the composite score created by averaging the z-scores of Selective Reminding Task, Face Name Task, and Visual Short Term Memory tasks.
Change in performance on executive function | At 3 months and at 9 months
  Change in performance on executive function will be measured using the composite score created by averaging the z-scores of Flanker Task, N-Back Task and Task Switch (fMRI task).
Change in brain function | At 3 months
  Change in resting state functional connectivity will be measured by resting State T2*weighted EPI-BOLD, a 10-minute task-free BOLD contrast sequence consisting of 300 volumes (TR=2000 ms/TE=30ms) at 3.4mm3 in-plane resolution and 3mm slice thickness. Participants will be instructed to keep their eyes open and maintain attention on a central gray fixation cross on a black screen.
Change in brain structure | At 3 months
  3D T1-Weighted multi-echo MPRAGE. Morphometric analyses will be based on this MRI sequence (not accelerated because the reliability of acceleration for multi-site studies has not yet been established). We will achieve spatial resolution of 1 x 1 x 1 mm voxels.
Change in task-related brain activation | At 3 months
  Change in functional connectivity and brain activation will be measured while performing Task Switch.
Change in functional performance | At 3 months and at 9 months
  Between-group magnitude of change in sum time of all tasks in the Timed Instrumental Activities of Daily Living (TIADL). Higher scores indicate greater impairment in functional performance.
Change in Depressive Symptoms | At 3 months and at 9 months
  Between-group magnitude of change in sum score using the self-report measure, Center for Epidemiologic Studies Depression Scale (CES-D). The scoring range is 0-60. Higher scores indicate the presence of more symptomatology.

OTHER OUTCOMES:
Change in Stress | At 3 months and at 9 months
  Between-group magnitude of change in sum score using the self-report measure, Perceived Stress Scale (PSS-10). The scoring range is 0-40. Higher scores indicate higher perceived stress.
Change in Self-Efficacy | At 3 months and at 9 months
  Between-group magnitude of change in sum score using the self-report measure, Self-Efficacy Survey. The scoring range is 10-40. Lower scores indicate lower self efficacy.
Change in Life Satisfaction | At 3 months and at 9 months
  Between-group magnitude of change in sum score using the self-report measure, Life Satisfaction Scale. The scoring range is 5-35. Lower scores indicate lower life satisfaction.
Change in Physical Activity | At 3 months
  Change in total score based on weekly self-report dairy about physical activity during training period.
Change in Diet | At 3 months
  Change in total score based on weekly self-report dairy about diet during training period.
Change in Social Activity | At 3 months
  Change in total score based on weekly self-report dairy about social activity during training period.
Change in Sleep | At 3 months
  Change in total score based on weekly self-report dairy about sleep during training period.
Change in Functional Abilities | At 3 months
  Change in total score based on weekly self-report dairy about functional abilities during training period.

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Kyu Lee, PhD, Principal Investigator — Posit Science Corporation
Locations (2):
- United States (2):
  - University of Iowa, Iowa City, Iowa
  - University of Texas at Dallas, Dallas, Texas

REFERENCES:
- [Derived] Lee HK, Basak C, Grant SJ, Ray NR, Skolasinska PA, Oehler C, Qin S, Sun A, Smith ET, Sherard GH, Rivera-Dompenciel A, Merzenich M, Voss MW. The Effects of Computerized Cognitive Training in Older Adults' Cognitive Performance and Biomarkers of Structural Brain Aging. J Gerontol B Psychol Sci Soc Sci. 2024 Jul 1;79(7):gbae075. doi: 10.1093/geronb/gbae075. PMID 38686621